CLINICAL TRIAL: NCT02637934
Title: Phase I Pilot Study of Biodistribution, Metabolism and Excretion of Novel Radiotracer [18F]Fluorthanatrace (FTT) by PET/CT
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 18815
Record Dates: First submitted 2015-12-18; First posted 2015-12-22 (Estimated); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Suspected Epithelial Ovarian, Fallopian Tube, or Primary Peritoneal Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Biodistribution (Experimental): The Biodistribution cohort will include up to 4 patients who will undergo a series of vertex to mid-thigh biodistribution [18F]FTT PET/CT scans over a period of approximately 4 hours.
  Up to 10 subjects were initially planned for this cohort, however, the first 4 subjects have been enrolled and initial data analysis for these completed. The decision was made to close enrollment for this cohort as we do not believe that we need to complete the up to 10 subjects originally planned for this cohort as the initial data shows consistent and repeatable data that we do not believe would change significantly with the addition of 6 more subjects.
  Interventions: Drug: [18F]FluorThanatrace; Radiation: PET/CT imaging sessions
- Dynamic (Experimental): The Dynamic cohort will include up to 36 patients who will undergo 1 static skull base to mid-thigh scans imaging post injection of [18F]FTT.
  Interventions: Drug: [18F]FluorThanatrace; Radiation: PET/CT imaging sessions

INTERVENTIONS:
Drug: [18F]FluorThanatrace
Radiation: PET/CT imaging sessions

SUMMARY:
Up to 40 evaluable women with known or suspected epithelial ovarian, fallopian tube, or primary peritoneal cancer will participate in two different imaging cohorts. The Biodistribution cohort will include up to 4 patients and the Dynamic cohort will include up to 36 patients. Human dosimetry will be calculated from the Biodistribution cohort. The Dynamic cohort date will evaluate preliminary information on uptake of [18F]FTT in gynecological cancer and compare with PARP-1 activity in tissue.

DETAILED DESCRIPTION:
Primary Objectives

• Evaluate PARP-1 activity in epithelial ovarian, fallopian tube, or primary peritoneal cancer using measures of uptake of [18F]FluorThanatrace

Secondary Objectives

* Evaluate the safety of [18F]FluorThanatrace
* Correlate [18F]FluorThanatrace uptake measures with BRCA mutation status
* Correlate [18F]FluorThanatrace uptake measures with PARP-1 activity in tumor.
* Determine biodistribution of the radioactive investigational drug ([18F]FluorThanatrace) in patients and calculate human dosimetry.
* Evaluate change in [18F]FluorThanatrace uptake measures after therapy

ELIGIBILITY:
Inclusion Criteria for Dynamic cohort

* Participants will be ≥ 18 years of age
* History of known or suspected epithelial ovarian, fallopian tube, or primary peritoneal cancer (may have primary or recurrent cancer at the time of study enrollment)
* At least one lesion ≥ 1.0 cm that is seen on standard imaging (e.g. CT, MRI, ultrasound, FDG PET/CT)

Exclusion Criteria for Dynamic cohort

* Females who are pregnant or breast feeding at the time of screening will not be eligible for this study; a urine pregnancy test will be performed in women of child-bearing potential at screening.
* Inability to tolerate imaging procedures in the opinion of an investigator or treating physician
* Any current medical condition, illness, or disorder as assessed by medical record review and/or self-reported that is considered by a physician investigator to be a condition that could compromise participant safety or successful participation in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2016-01-14 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Number of Adverse Events | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Fiona Simpkins, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Makvandi M, Pantel A, Schwartz L, Schubert E, Xu K, Hsieh CJ, Hou C, Kim H, Weng CC, Winters H, Doot R, Farwell MD, Pryma DA, Greenberg RA, Mankoff DA, Simpkins F, Mach RH, Lin LL. A PET imaging agent for evaluating PARP-1 expression in ovarian cancer. J Clin Invest. 2018 May 1;128(5):2116-2126. doi: 10.1172/JCI97992. Epub 2018 Apr 16. PMID 29509546